CLINICAL TRIAL: NCT02283749
Title: BrUOG L301: Xofigo Following Frontline-Line Chemotherapy For Patients With Non-Small Cell Lung Cancer and Bone Metastases
Brief Title: BrUOG L301 With Non-Small Cell Lung Cancer and Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angela Taber MD (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Angela Taber MD, Principal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 301
Record Dates: First submitted 2014-10-30; First posted 2014-11-05 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer With Bone Metastatses
Keywords: NCSLC; lung cancer; non small cell lung cancer; bone metastases; maintenance
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Xofigo (Experimental): Xofigo, 50 kBq/kg body weight, will be administered in the nuclear medicine department as a bolus intravenous (IV) injection (up to 1 minute) at intervals of every 4 weeks for up to 6 cycles.
  Interventions: Biological: Xofigo

INTERVENTIONS:
Biological: Xofigo — This is a radio-isotope
  Other Names: Radium -223

SUMMARY:
In this study patient's will receive the medicine Xofigo which is a radioactive drug that is FDA approved to treat prostate cancer that has spread to the bones. Xofigo has not previously been tested to treat lung cancer that has spread to the bones. Your doctors are studying the effects, good and bad, of Xofigo when used to treat lung cancer that has spread to the bones.

DETAILED DESCRIPTION:
In this study patient's will receive the medicine Xofigo which is a radioactive drug that is FDA approved to treat prostate cancer that has spread to the bones. Xofigo has not previously been tested to treat lung cancer that has spread to the bones. Your doctors are studying the effects, good and bad, of Xofigo when used to treat lung cancer that has spread to the bones. Your doctors will also be evaluating changes in health related quality of life using the EORC QL-C20 and QOL-BM22 questionnaires. They will also evaluate the impact of treatment on the Alkaline phosphate levels (by way of lab draws) in patients and measure the progression free survival and overall survival of patients with stable or responding disease after the front line chemotherapy treated with Xofigo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Advanced non-small cell lung cancer with bone metastases.
* Stable or responding disease after completion of initial systemic chemotherapy as defined by RECIST criteria. Site to submit confirmation to BrUOG.
* At least 3 weeks must have elapsed since completion of last chemotherapy and 4 weeks since last radiation, prior to first dose of Xofigo. Patients are not permitted to receive any form of 'maintenance' chemotherapy or biologic/targeted anticancer therapy while being treated on this study
* Life expectancy of at least 12 weeks (3 months).
* Patients with treated brain metastases are allowed, but must have brain imaging showing evidence of stability since most recent treatment for brain mets, prior to first dose of Xofigo. For patients with brain metastases only, brain imaging is required. Patients who do not have brain metastases or symptoms of potential brain metastases are not required to have baseline brain imaging, but this must be confirmed in writing
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1.
* Required entry laboratory parameters within 14 days of study entry: White Blood Cell Count (WBC) ≥ 3,000/mm3; Absolute Neutrophil Count (ANC) ≥ 1,500/mm3; Platelet (PLT) count ≥ 100,000/mm3; Hemoglobin (Hgb) > 9g/dl, Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN ; Creatinine ≤ 1.5 x ULN; Albumin > 2.5 g/dL.
* Concurrent treatment with bisphosphonates and denosumab is allowed. Information on start and stop date and drug with dose to be sent to BrUOG if patient to be treated concurrently.
* Prior skeletal related events (pathologic fracture, radiation or surgery to bone, or spinal cord compression) are allowed if they have been managed and now patient is stable for 4 weeks prior to study entry. Must submit how events managed to BrUOG for documentation to confirm eligibility criterion. (For example, if a patient experienced a SSE and had radiation for 2 weeks they must then be stable for 4 weeks after the completion of radiation prior to study entry)
* Subjects must be able to understand and be willing to sign the written informed consent form.
* All acute toxic effects related to prior treatment(s) must have resolved to NCI-CTCAE v4 Grade 1 or less at the time of signing the Informed Consent Form (ICF) except for alopecia.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the treating physician.
* Willing and able to comply with the protocol, including follow-up visits and examinations

Exclusion Criteria:

* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Radium Ra 223 dichloride) for the treatment of bony metastases
* No prior invasive malignancy within the prior two years. However, patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer or asymptomatic prostate cancer) are eligible
* Untreated brain metastases.
* Any other serious illness or medical condition that in the investigator's opinion would interfere with protocol treatment, such as but not limited to: Any active infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4 Grade 2: Cardiac failure New York Heart Association (NYHA) III or IV
* Women who are pregnant or breast-feeding.
* Inability to comply with the protocol and/or not willing or who will not be available for follow-up assessments.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than Ra 223 dichloride.
* Major surgery within 28 days of starting study drug. Central venous catheter placement is not considered major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-05 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (1):
- Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xofigo
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Xofigo
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 58 [44 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Skeletal Events (SSE) in Patients Receiving Xofigo With NSCLC and Bone Metastases
Description: Number of Participants with Symptomatic Skeletal Events (SSE) Receiving Xofigo With NSCLC and Bone Metastases
Time Frame: Approximately every 2 months for up to a year
Measure: Number; unit: Number of participants experiencing SSE
Arm/Group | Xofigo
Number analyzed (Participants) | 5
Number of participants experiencing SSE | 1

2. Secondary Outcome: Progression-free Survival of Patients With NSCLC and Bone Metastases and Stable or Responding Disease After Front-line Chemotherapy Treated With Xofigo
Description: To measure progression-free survival of patients with NSCLC and bone metastases and stable or responding disease after front-line chemotherapy treated with Xofigo. Post 1 year of follow up the number of patients that remain stable or responding
Time Frame: During treatment (6 cycles, 1 cycle=4 weeks) and through 1 year post treatment
Population: Post 1 year of follow up the number of patients that remain stable or responding
Measure: Count of Participants; unit: Participants
Arm/Group | Xofigo
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Overall Survival of Patients With NSCLC and Bone Metastases and Stable or Responding Disease After Front-line Chemotherapy Treated With Xofigo
Description: To measure overall survival of patients with NSCLC and bone metastases and stable or responding disease after front-line chemotherapy treated with Xofigo
Time Frame: During treatment (6 cycles, 1 cycle=4 weeks) and through 1 year post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Xofigo
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Any serious adverse event occurring after the patient has provided informed consent and until 4 weeks (30 days +1 week) after the patient has stopped study participation must be reported.
Description: Any adverse event occurring after the patient has provided informed consent and until 4 weeks (30 days +1 week) after the patient has stopped study participation were captured.
Arm/Group | Xofigo
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Xofigo (N=5)
Albumin (hypo) (Investigations) | 1 (1)
ANC (Investigations) | 1 (1)
Anorexia (Investigations) | 1 (1)
Bilateral Leg Cramps (Investigations) | 1 (1)
Dehydration (Investigations) | 2 (2)
Diarrhea (Investigations) | 1 (1)
Dizziness (Investigations) | 2 (2)
Eye disorder other ( kaleidoscope vision) (Investigations) | 1 (1)
Fatigue (Investigations) | 1 (1)
flatulence (Investigations) | 1 (1)
HGB (Investigations) | 3 (3)
HTN (Investigations) | 3 (3)
Insomnia (Investigations) | 1 (1)
Lymph (Investigations) | 3 (3)
Menorrhagia (Investigations) | 1/1 (1)
NA (hypo) (Investigations) | 1 (1)
nausea (Investigations) | 3 (3)
Oral Hemorrhage (Investigations) | 1 (1)
Pain (back, R hip, Ribs ) (Investigations) | 1 (1)
PLT (Investigations) | 2 (2)
WBC (Investigations) | 1 (1)
weight gain (Investigations) | 1 (1)
Dyspnea (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02283749/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02283749/SAP_001.pdf